CLINICAL TRIAL: NCT01041599
Title: Assessment of the Association Between Albuminuria and Arterial Stiffness in Diabetic Patients, Hypertensive Patients and Healthy Controls
Brief Title: Correlation of Albuminuria With Arterial Stiffness
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fatih Tufan, assoc prof MD, Istanbul University
Other Study IDs: 4154
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus; Hypertension; Albuminuria; Vascular Stiffness
Keywords: Diabetes Mellitus; Hypertension; Albuminuria; vascular stiffness
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Albuminuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetic patients: Hypertensive and normotensive patients with type 2 diabetes mellitus
- Hypertensive patients: Patients with essential hypertension
- Healthy subjects: Healthy subjects

SUMMARY:
The investigators aim to investigate the relationship between albuminuria and arterial stiffness in diabetic patients, hypertensive patients and healthy subjects.

DETAILED DESCRIPTION:
CONTEXT: Albuminuria is an important cardiovascular risk factor. Arterial stiffness also gives important information about atherosclerosis. Oscillometric methods may be useful in assessing arterial stiffness in a mainly operator independent way.

OBJECTIVE: We aim to investigate the relationship between albuminuria and arterial stiffness measured with an oscillometric device in diabetic patients, hypertensive patients and healthy subjects.

METHODS: 152 diabetic patients, 152 hypertensive patients and 152 healthy subjects are planned to be enrolled in this study. The measurements will be done between 9:00 and 13:00. After the measurements, blood and urine samples will be obtained, centrifugated and kept in -80°C until assayed. Afterwards, echocardiographic left ventricle mass index will be calculated. The correlation between albuminuria and arterial stiffness will be assessed as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus
* Hypertension
* Healthy subjects

Exclusion Criteria:

* Symptomatic cardiovascular diseases (heart failure, history of myocardial infarction, etc.)
* Renal failure
* Pregnancy
* Diseases of the aorta

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes, patients with hypertension and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Correlation between albuminuria and arterial stiffness | Albuminuria and arterial stiffness will be assessed simultaneously (i.e. in the same morning)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kaya, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Abdullah Ozkok, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Bahtiyar Toz, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Kadri Atay, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Hamza Ugur Bozbey, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Ercan Bicakci, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Mehmet Besiroglu, MD, Study Chair — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine; Fatih Tufan, MD, Study Director — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine Division of Geriatrics; Tevfik Ecder, Prof, Principal Investigator — Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine Division of Nephrology; Miklos Illyes, MD, Ph. D, Study Director — Heart Institute, Pecs University Faculty of Medicine, Pecs/Hungary; Kamil Nas, MD, Study Director — Szent Janos Hospital Radiology Department, Budapest/Hungary; Molnar Ferenc, Study Director — Tensiomed Arterial Stiffness Centre, Budapest/Hungary
Locations (1):
- Istanbul Univesity Istanbul Medical Faculty Department of Internal Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
yes